CLINICAL TRIAL: NCT01524081
Title: Phase 3 Study of Antibiotic Prophylaxis Use Prior Emergent Surgery, Because of Acute Appendicitis
Brief Title: Antibiotic Prophylaxis in the Prevention of Surgical Site Infections After Selected Urgent Abdominal Surgical Procedures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Faculty Hospital Na Bulovce (Other)
Responsible Party: Principal Investigator, Zuzana Serclova, MD, Head of ICU - Department of Surgery, Principal Investigator, The Faculty Hospital Na Bulovce
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FNB_ATB
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-01

CONDITIONS: Acute Appendicitis; Perforated Gastroduodenal Ulcer; Small Bowel Obstruction
Keywords: antibiotic prophylaxis; emergent surgery; surgical site infection
MeSH Terms: conditions — Appendicitis; Surgical Wound Infection | interventions — Metronidazole; Cefuroxime; Benchmarking; Amoxicillin; Clavulanic Acid; Fluconazole; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (6):
- APPE - antibiotic prophylaxis (Experimental): Patients indicated for emergent appendectomy with antibiotic prophylaxis
  Interventions: Drug: Metronidazole, Cefuroxime
- GERD - antibiotic prophylaxis (Experimental): Patients indicated for emergent surgery due to gastroduodenal perforation with antibiotic prophylaxis.
  Interventions: Drug: Amoxicillin (+ clavulanic acid) and Fluconazole
- ILEUS - antibiotic prophylaxis (Experimental): Patients indicated for emergent due to small bowel obstruction with antibiotic prophylaxis
  Interventions: Drug: Metronidazole, Cefuroxime
- APPE - placebo (Placebo Comparator): Patients indicated for emergent appendectomy without antibiotic prophylaxis. Placebo (saline) was administrated.
  Interventions: Drug: Placebo
- GERD - placebo (Placebo Comparator): Patients indicated for emergent surgery due to gastroduodenal perforation without antibiotic prophylaxis. Placebo (saline) was administrated.
  Interventions: Drug: Placebo
- ILEUS - placebo (Placebo Comparator): Patients indicated for emergent due to small bowel obstruction without antibiotic prophylaxis. Placebo (saline) was administrated.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metronidazole, Cefuroxime — administration of Cefuroxime 1.5 g and Metronidazole 1g in 2 following intravenous infusions 60 minutes prior the surgery.
  1. - Cefuroxime in 100ml saline
  2. - Metronidazole in 500ml saline
  Other Names: Zinacef 750mg (Cefuroxime 750mg, Glaxo Group Ltd., UK); Metronidazol 500mg (Metronidazole 500mg; B.Braun Melsungen AG, Germany)
  Arms: APPE - antibiotic prophylaxis; ILEUS - antibiotic prophylaxis
Drug: Amoxicillin (+ clavulanic acid) and Fluconazole — Administration of amoxicillin (+ clavulanic acid) 2.4 g and Fluconazole 800mg in 2 following intravenous infusions 60 minutes prior the surgery.
  1. - 2x amoxicillin in 100ml saline
  2. - Fluconazole in 500ml saline
  Other Names: Amiksiklav 1,2 g (amoxicillinum natricum 1000mg, acidum clavulanicum 200mg; Lek Pharmaceuticals d.d., Ljubljana, Slovenia; Fluconazol 200ml (fluconazolum 400mg; Baxter; Czech Republic)
  Arms: GERD - antibiotic prophylaxis
Drug: Placebo — Administration of saline infusion (Natrii chloridum: 9,0 g/l) 60 minutes prior the surgery
  1. - 100ml saline solution
  2. - 500ml saline solution
  Other Names: F1/1 (saline solution; 0,9% NaCl; Baxter Czech Republic)
  Arms: APPE - placebo; ILEUS - placebo
Drug: Placebo — Administration of saline infusion (Natrii chloridum: 9,0 g/l) 60 minutes prior the surgery
  1. - 2x 100ml saline solution
  2. - 500ml saline solution
  Other Names: F1/1 (saline solution; 0,9% NaCl; Baxter Czech Republic)
  Arms: GERD - placebo

SUMMARY:
Aim of prospective randomized a placebo controlled study is to prove that in case of acute surgical procedure due to appendicitis, ileus of small bowel and perforation of small bowel and stomach appropriately administered antibiotic prophylaxis is effective with lower incidence of infection in surgical site and comparable risk of development of other nosocomial infections versus group without antibiotic prophylaxis. Secondary aim is to determine risk of developing nosocomial infection in the above mentioned group of patients, identify group of patients which does not benefit from prophylaxis, and compile financial costs for antibiotic prophylaxis and treatment of nosocomial infections and thus the background for the recommended procedure with regards that such prospective study does not exist in the Czech Republic.

DETAILED DESCRIPTION:
Introduction Infection related to surgical procedure was always considered the main cause of mortality end morbidity in surgical patients. ATB prophylaxis has become the breakthrough in surgical praxis in terms of prevention of surgical postoperative complications (Surgical Site Infection - SSI) and radical improvement of surgical results. ATB prophylaxis prior to intervention procedures presents however 1/3 of costs for medicinal products and it is also potentially hazardous. Even single use of antibiotic agent can be a cause for development of nosocomial infection with indispensable mortality and costly treatment. Several recommendation in worldwide literature have been presented during the last 10 years which concerned indications and route of administration of antibiotics prior to scheduled or acute surgical procedure; indications for acute procedures broaden and it increases the consumption of antibiotics. Excessive pre-hospital and hospital exposure to antibiotics is however related to development of microbial resistance which shows in higher incidence of nosocomial infections (health care - associated infection - HAI) - urinary infections, pneumonia, catheter infection and another diseases such as Clostridium colitis caused by highly virulent type. Moreover some studies suggest bad compliance in dosing and timing of antibiotic prophylaxis which causes only the negative effect of prophylaxis without positive affection of SSI. This knowledge and disagreement led us to elaboration of protocol for prospective randomized placebo controlled study which could be the base for correct surgical praxis in investigator's conditions.

Aim of the project The aim of this prospective randomized placebo controlled study is to prove the positive effect of antibiotic prophylaxis on the incidence of SSI in patients with comparable risk of developing other nosocomial infections in case of acute abdominal procedures for diagnosis such as appendicitis, ileus of small bowel and stomach or small bowel perforation and thus with exclusion of tertiary peritonitis. Secondary aim is to identify the group of patients in which risk of developing nosocomial infection exceeds benefit of ATB prophylaxis. Tertiary aim is to assess whether preoperative microbial screening has its significance for reduction of HAI. After comparing the financial cost of therapy (including SSI and HAI generally) it will be possible to submit background for proposal of recommended procedure for administration of antibiotic prophylaxis in the most common acute surgical procedures with regard to risk factors for genesis of nosocomial infections. Such prospective randomized placebo controlled study has not been conducted in the Czech Republic; further study with similar target group of patients (very common in surgical praxis) has not been published in world literature.

Hypothesis Correctly administered antibiotic prophylaxis prior to acute abdominal procedures reduces frequency of SSI. It can increase the frequency of severe nosocomial infections in risk group of patients. rational use of antibiotic prophylaxis should however lead to reduction of incidence of nosocomial infections with clinical and socioeconomic impacts including prevention of feared severe infections associated with health care (HAI).

Methodology

Method is aimed at:

1. Assessing the effect of risks to development of nosocomial infections on behalf of patient (ASA, morbidity, relevance of the actual disease, microbial screening targeted on community infection, BMI, previous hospitalization in health care facility).
2. Assessing perioperative influence on the genesis of nosocomial infections (correct administration of ATB prophylaxis- protocol control, perioperative influences - blood loss, body temperature, extend of inflammation, SIRS sings, duration of surgery, ICU stay, microbial profile, analgesia, physiotherapy, complications assessment).
3. Assessing the influence of ATB if those are correctly administered on the genesis of SSI in acute procedures (length of hospitalization, length of treatment and complications).
4. Long term and socioeconomic impacts of SSI (60 days follow up, life quality assessment), standard proposal. After completion of patient monitoring the analysis of cost for hospitalization including medication, surgery and postoperative outpatient control will be conducted using the hospital information system.

Appropriate patients to be enrolled in the study are all patients with following diagnosis operated at the site: Acute appendicitis (classical or laparoscopy appendectomy), ileus of the small bowel (adhesiolysis, enterotomy with suction or resection of small bowel), perforated stomach or duodenal ulcer (classical excision of the ulcer and suture of the GIT wall), i.e. patients without stercoral peritonitis. Patient will be definitely included if they signed the preoperative informed consent form which they were able to understand well and whose diagnosis was confirmed during surgery. Patients will be excluded if they are younger than 18 years of age, pregnant females, and patients with known allergy to administered ATB and also if their mental state does not allow appropriate instruction and signing of the informed consent and further patients who used ATB in the course of last 2 weeks.

Preoperative care, actual surgical procedure and subsequent postoperative care are not the direct subject of study and will be conducted according to so far known procedures.

Patient will be administered therapeutic agent (antibiotic) or placebo in form of intravenous infusion 60 minutes prior the surgical procedure due to suspicion of the above mentioned diagnosis. If the surgery lasts for more than 3 hours, the infusion will be repeated. After analysis of the most common pathogens in individual clinical diagnosis, microbiologist chose following preparations: Acute appendicitis - Cefuroxim (Zinacef 1.5 g) + Ornidazol (Avrazor 1g), perforated ulcer - Aminopenicillin + inhibitor (Amoksiklav 2.4 g) + Fluconazole 800mg i.v., ileus of small bowel - Cefuroxim (Zinacef 1.5 g) + Metronidazol (Avrazor 1g). Surgeon will confirm the definite diagnosis during surgery which will confirm the definite inclusion in the study. Surgeon will not be present dilution or administration of the agent. Nobody from patient's attending study personnel will not be able to distinguish whether the patient was administered antibiotic or saline solution. The prophylaxis will be extended for 24 hours in common half-dosage according to publication sources.

Randomization will be conducted using generator of random numbers. This sequence will be incorporated in simple digital patient database internet access to which will be password protected. One educated ICU nurse will enter only basic patients´ data and system itself will determine whether to prepare placebo or diluted antibiotic. Since that moment this information will be confidential and software will be accessible only for entering other monitored parameters. Dividing into individual groups will be conducted in interim controls after six months intervals and final division after completion of study. Totally there will be 2 major groups and 6 subgroups and those 3 subgroups according to individual diagnosis each one with 1 control group. If severe complication (allergy reaction) occurs, the principle investigator can uncover the blinding using specific password; system entry will automatically mean exclusion of the patient from study.

Patients will be discharge from the hospital based on criteria (agreement of the patient, without signs of severe infection (SIRS), sufficient oral intake, sufficient analgesia with oral analgesics, would treatable in the outpatient department); patient will be treated as outpatients in case of complications; patients will be questioned on the phone in case of uncomplicated course and they will be ask to fill out life quality questionnaire (SF36) on the day 30 and 60.

Demographic data on included patient and monitored data will be recorded into special cards and transmitted in the specifically created software to further processing.

Investigators assume to include total of 500 patients during 3 years.

Time schedule:

1. year of the project: creation of the randomization program, personnel education, software creation, inclusion of 130 patients with appendicitis diagnosis, 18 patients with ileus of small bowel and 35 patients with perforation of ulcerous disease. Data processing. Results will be evaluated at the end of the year.
2. year of the project: Inclusion of 130 patients with appendicitis diagnosis, 18 patients with ileus of small bowel and 35 patients with perforation of ulcerous disease. Data analysis will be performed and subgroup analysis and partial results will be processed and presented.
3. year of the project: Inclusion of 90 patients with appendicitis diagnosis, 14 patients with ileus of small bowel and 30 patients with perforation of ulcerous disease. Follow up termination. Definite data collection, analysis, results evaluation including financial analysis. Standard proposal. Presentation in national and international forums, publications.

Principle investigator will apply the created protocol and will continuously control its compliance including schedule, will process interim data, will evaluate data compliance with literature and will prepare their presentation and publication and will process final results. 2nd co-worker is guarantees the microbiological part of the project; 3rd and 4th co-workers will collect rather large amount of data and will enter them in created system. 5th and 6th co-workers will control including appropriate patients in study (it means acute procedure), % of included patients out of number of suitable patients is an important criterion for significance of gathered data. They also cooperate in presentation data processing. 7th co-worker controls correctness of data collection. 5 specifically educated independent nurses who do not attend the patient (24 hour service) will prepare infusions for patients according to acquired randomization data - placebo or monitored group. Administrative worker will select data from the information system and patients´ files, file and selects study cards and supervises their correct completion.

Means of data collection Data collection will be conducted in terms of preoperative examination: Demographic data (age, diagnosis, co-morbidity expressed by score - ASA, BMI, blood count, CRP), microbiology samples for detection of influence of community pathogens, especially presence of multiresistant pathogens - Clostridium difficile will be sought.

In course of surgery: evaluation of perioperative finding, SSI risk 0-3 point; contamination scoring I-IV, body temperature monitoring (BT), blood loss (including weighing of screens), length of surgery.

In postoperative period will be recorded: number of transfusion preparations, number of days on UPV, days at ICU, oral intake, physiotherapy, invasive inlets (peripheral venous catheter, permanent urinary catheter, nasogastric tube, drains) and quality of analgesia (Visual Analog Scale - VAS).

On discharge: samples collection for microbiological examination, record of SSI incidence and other HAI defined according to criteria of National Healthcare Safety Network (NHSN), completion of assessment of life quality questionnaire (SF36).

After discharge: complications will be recorded till day 30 and 60 (SSI and HAI), life quality assessment. After completion of patient monitoring the analysis of cost for hospitalization including medication, surgery and postoperative outpatient control will be conducted using the hospital information system.

Statistics:

Morbidity which ranges from 15 to 20%, investigators consider 10% as clinically significant reduction. Minimal extent of each collection is 118 when considering 5% level of significance for single sided test and test power 70%; minimal extent of each collection for portion of nosocomial infection 6-10% is 234 in case of clinically significant decrease by 5%. Estimates of numbers required for detection of clinical difference of two days (standard deviation estimate 2.6 for appendicitis respectively 3.2 for perforation and 2.3 for ileus of small bowel) lead to values 36, 47 a 25 people in each group. Total number for each set is 250 people and it fulfills the above mention criteria and ranges 175, 50 and 25 in each subgroup are sufficient. Group homogeneity will be compared based on descriptive statistical methods; risk factors will be evaluated using regression analysis and multivariant analysis. When comparing basic factors p<0.05 will be considered as clinically significant in case of above given test power.

Patient informed consent (short version, complete version was approved by ethics committee and is enclosed in appendix): Study description: Each surgical procedure has its own risk so called postoperative infectious complications. One possibility how to prevent those complications is the preventive administration of antibiotics just prior the procedure - so called antibiotic (ATB) prophylaxis. There is no clear evidence for positive effect of ATB prophylactic use in some acute surgical procedures. On the other hand introduction of ATB prophylaxis has its complications. Aim of study: Aim of the study is the recommendation whether in given cases administration of ATB prophylaxis has positive effect on reduction of incidence of postoperative infectious complications and whether this benefit is higher than risks related to ATB administration. Inclusion in study and conductance: Single inclusion is only based on the decision of patient (approximately 500 patients). Study participation will be offered to patients who will be operated on due to acute appendicitis, perforated stomach or duodenal ulcer or due to ileus of small bowel. Pregnant and lactating females are excluded from the study. After patient's consent with study participation the intravenous preparation will be administered which contains active substance (antibiotic) or placebo (only saline solution). Both administered substances are registered preparations administered for given purpose in general praxis. The chance of application of either active preparation and or placebo is 50:50. Patient will be telephonically inquired about concrete postoperative complications on day 30 and 60 after surgery. If there is suspicion on complication, patient will be examined and treated using standard procedure. He will be further asked for completion of questionnaire about life quality. Health risks: This study is not related to practically any excessive risk. ATB and placebo administration does not in any way influence the surgical procedure or postoperative care. Non-invasive sample collection for cultivation (urine collection, sputum collection -secretion from respiratory tract mucosa, smear from throat and stool). Compensation for bodily harm: If patient obliges to study physician's instructions and her/his team and health damage of patient occurs as a result of administration of any preparation, the study sponsor will cover all cost for treatment of this damage which is not covered by patient's health insurance. Patient's declaration: I, undersigned, agree with my participation in study. I am older than 18 years of age. I was informed in detail about the aim of study, its procedures and what it is expected from me. Study physician explained me the expected benefits and possible health risks. I acknowledge that conducted study is an investigation activity. Study is randomized and therefore I acknowledge possibility of random assignment into individual groups which differ in therapy. I fully understood and I have the opportunity to ask additional questions which were satisfactory answered to me. I informed study conducting physician about all my diseases and medications which I have been taking over the last 28 days and also about medication which I currently take. I declare that I do know that I am pregnant at time of inclusion in the study. I understood that I can discontinue or withdraw my participation in the study at any time without affecting course of my further treatment. My personal data will be kept in full confidentiality after study enrollment according to applicable laws in the Czech Republic. Based on my given consent my original medical information could be accessed to authorized acquired data by sponsor representatives, independent ethics committees and international or local competent authorities (The State Institute for Drug Control in the Czech Republic). Confidentiality protection of personal data is guaranteed for those cases. There will not be any cost to me for my participation in study and concomitantly study enrollment is not related to any financial reward. I understood that my name will never be present in reports about this study. (date, name, signature) Cooperation Working site of co-worker participates in postgraduate education; co-worker is recognized surgical expert and therefore he is guarantee for correct study conductance and results applications in praxis; the cooperation will be confirmed by agreement.

Discussion Investigator's working site will conduct internal retrospective study dealing with SSI in patients with appendicitis and stomach ulcer perforation. 180-200 acute appendectomies will be performed every year with SSI frequency 2.5 - 18.5% according to contamination. Group of patient with stomach ulcer perforation will be evaluated similarly (n=42) with SSI 14.3%, total morbidity 35% and mortality 11.9%. All of those data correlate with results from the world literature however it is possible that after retrospective assessment correct monitoring of ATB prophylaxis (40% compliance) and patient stratification will reduce the frequency of complications.

Information Working site of designer performs hundreds of the above given operations which a presumption for completion of the study aims. Especially young surgeon will participate in this study who will manage methodology of hospital care as well as surgery under supervision of experienced physician and will educated for patients´ monitoring. Statistical evaluation will be performed by professional statistician. Principle investigator has numerous experiences with clinical studies and she/she published his/her results in journals. Other specific equipment is not necessary for study procedure.

Conclusion Proposed prospective randomized double blinded study will provide clear results assessing effect of administration of ATB prophylaxis on the incidence of SSI and other HAI in case of the most common acutely performed surgical procedures. Risk factor analysis and costs for treatment will aid to determine group of patients who will benefit from prophylaxis and vice versa.

Expected results and significance of the project Project results will be used as background for establishing recommended procedure of antibiotic prophylaxis administration in surgery. Standardized protocol will be introduced for patients monitoring including monitorzation of nosocomial infections which is can be applied in general surgical praxis. Simple universal software will be created in terms of study which manages patient database and thus enables rapid concurrent assessment of health care quality. Respective reduction of nosocomial infections frequency should result in significant economic benefit for surgical praxis. With regard that similar complex prospective study has not been published in national and international magazines, publication in impact journal; socioeconomic analysis will be published especially in national medical journals so it would be easily accessible.

Project should aid the prevention of nosocomial infections (HAI) and reduction of their genesis and thus to increase surgical care, shorten hospitalization and should have impact on the whole society.

ELIGIBILITY:
Inclusion Criteria:

* patient older > 18 years
* Patient indicated for emergent surgery for:

acute appendicitis / perforated gastric or duodenal ulcer / small bowel obstruction

* The patient can understand the aim of the study and sign informed consent (including language barriers)
* The diagnose is confirmed intraoperatively

Exclusion Criteria:

* Refused the participation in the study and
* uninsured self-payers
* Patients with known allergy to the substance administered during the study or chronic medication contraindicated with study drug
* Pregnant or breastfeeding women
* Use of antibiotics in the last 2 weeks
* Known serious illness (heart failure, renal failure, liver failure, CNS disorders)
* Signs of infectious mononucleosis and risk of infectious endocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2008-07; Primary Completion 2011-07 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Surgical Site Infection rate | 30 days after surgery
  The evidence of Surgical Site Infection (SSI) using clinical definition CDC/NHSN)

SECONDARY OUTCOMES:
Hospital Acquired Infection /HAI/ | 60 days after surgery
  Incidence of HAIs during the 60 days after surgery. Diagnosis confirmed using criteria CDC/NHSN

CONTACTS AND LOCATIONS:
Overall Officials: Ondrej Ryska, MD, Principal Investigator — Department of surgical, Faculty Hospital Bulovka, Prague, Czech Republic
Locations (1):
- Faculty Hospital Bulovka, Prague, Czechia